CLINICAL TRIAL: NCT06303778
Title: Combining a Smartphone App With Medications to Manage Heavy Drinking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 22-141; HX003742-01A1 (Other Grant/Funding Number: VA HSR&D)
Record Dates: First submitted 2024-02-09; First posted 2024-03-12 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: alcohol use disorder; substance use disorder; medications for AUD; smartphone app; primary care; mobile health
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Following completion of informed consent and baseline assessments, participants will be randomized in a 1:1 ratio to MAUD+SD-App or MAUD only conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (Active Comparator): Participants assigned to the standard care condition will receive standard MAUD care delivered by their CPSs and will not receive access to SD-App. Three medications, naltrexone, disulfiram, and acamprosate, have been approved by the Federal Drug Administration and topiramate has been recommended by the VA/DoD clinical practice guidelines for SUD. MAUD includes these four medications. All medication decisions will be between the CPS and the Veteran and not influenced by study participation.
  Interventions: Other: Standard Care
- Combined MAUD+SD-App (Experimental): In addition to standard MAUD care, participants assigned to the MAUD+SD-App condition will receive access to the Stand Down app at randomization.
  Interventions: Other: Stand Down mobile app

INTERVENTIONS:
Other: Stand Down mobile app — The Stand Down mobile app is a smartphone-based stand-alone intervention designed to help persons manage drinking and alcohol-related problems on their own. The app is based on principles of motivational enhancement and cognitive-behavioral therapies and comprises 7 modules organized around 4 goals: (i) Enhance awareness of drinking patterns (assessment and personalized feedback), (ii) Establish and monitor progress towards drinking goal - i.e., moderation or abstinence, (iii) Manage cravings and other problems using in-the-moment tools, and (iv) Connect users with other types of support.
  Arms: Combined MAUD+SD-App
Other: Standard Care — Participants assigned to the standard care condition will receive standard MAUD care delivered by their CPSs and will not receive access to SD-App. Three medications, naltrexone, disulfiram, and acamprosate, have been approved by the Federal Drug Administration and topiramate has been recommended by the VA/DoD clinical practice guidelines for SUD. MAUD includes these four medications. All medication decisions will be between the CPS and the Veteran and not influenced by study participation.
  Arms: Standard Care

SUMMARY:
One in 10 Veterans have an alcohol use disorder. However, few Veterans receive evidenced-based psychosocial interventions or medications to treat alcohol use disorder. Barriers to receiving these treatments include long wait times, stigma, and long distances from treatment facilities. Even fewer Veterans receive psychosocial and medication interventions together, despite clinical practice guidelines recommending both and evidence of better outcomes. Expanding access to these treatments in primary care is a VA priority but delivering psychosocial interventions is difficult in this setting, and medication is often the only option. Smartphone apps that deliver alcohol interventions may improve drinking outcomes and ensure Veterans can receive both treatments in primary care. This study will determine whether medications and an app for alcohol use problems offered to Veterans in primary care results in improved drinking outcomes, compared to Veterans receiving medications only. Study data will inform how to spread the app across the VA nationally.

DETAILED DESCRIPTION:
Background: Alcohol use disorder (AUD) affects 1 in 10 Veterans and is associated with significant morbidity and mortality. However, few individuals receive evidenced-based psychosocial interventions or medications for AUD (MAUD). Common barriers to treatment include long wait times, stigma, and distance from treatment facilities. Despite clinical guidelines and evidence indicating superior outcomes, even fewer individuals receive MAUD and psychosocial interventions conjointly. The VA prioritizes expanding access to AUD interventions in primary care, but it is difficult to deliver psychosocial interventions in primary care, and care often includes MAUD only. Smartphone mobile applications (apps) that deliver psychosocial interventions concurrent with MAUD may address the gap between recommended and current practices for AUD and appeal to Veterans who prefer to receive their AUD care in primary care. Alcohol intervention apps have been associated with improved drinking-related and mental health outcomes. Self-monitoring of alcohol use, a common feature in apps, may also increase MAUD adherence. Step Away, an app for self-management of alcohol use problems, is designed to guide development and use of personalized strategies to moderate or abstain from drinking. In single-arm cohort studies, the investigators assessed the acceptability and usability of Step Away and Stand Down (SD-App), the Veteran version of the app and focus of this proposal, among Veterans with alcohol use problems. The apps received favorable ratings regarding perceived effectiveness, efficiency, and overall satisfaction, and were associated with reductions in heavy drinking days and drinking-related consequences.

Significance: This study has the potential to substantially improve Veterans' receipt of guideline-concordant AUD care and support national VA initiatives to increase access to AUD care in general healthcare clinics.

Innovation & Impact: To the investigators' knowledge, no prior study has evaluated the effectiveness of an alcohol-related intervention, delivered by smartphone, with MAUD in primary care. Smartphone apps can be scaled up at relatively low cost, potentially saving lives and improving the quality of care of tens of thousands of Veterans.

Specific Aims: The two aims are to: 1) determine whether MAUD plus SD-App offered to primary care patients diagnosed with AUD, compared to MAUD only, results in (a) greater reductions in heavy drinking days, from baseline to 6-months (primary), (b) greater improvements in alcohol consequences, alcohol use risk levels, and mental health outcomes, from baseline to 6-months (secondary), 2) conduct a process evaluation to identify factors that influence the adoption, implementation, and sustainability of SD-App in combination with MAUD in VA primary care from Veterans', clinical pharmacist specialists' and clinical leaders' perspectives. The investigators will also explore whether MAUD plus SD-App increases MAUD 6-month adherence relative to SD-App alone.

Methodology: Guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance framework, this Hybrid 1 effectiveness-implementation trial will enroll 330 Veterans across 15 VA sites. Veterans between ages 18-80, meeting AUD criteria, and planning to initiate MAUD will be randomized to MAUD+SD-App or MAUD only. Participants randomized to MAUD+SD-App will receive access to SD-App. MAUD will be prescribed by VA clinical prescribers per standard care. The primary and secondary outcomes will be assessed at baseline, 3-, 6- and 12-months using participant self-report and electronic medical record data. The investigators will complete qualitative interviews to assess Veterans', clinical pharmacists', and clinical leaders' perspectives on barriers and facilitators to adoption, implementation, and sustainability of SD-App in combination with MAUD in primary care.

Next Steps/Implementation: If MAUD+SD-App improves drinking outcomes, the investigators will work closely with the operations partners to review study findings and to develop a tailored implementation strategy to support widespread implementation across VA primary care.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, Veterans must be:

* 1) diagnosed with an AUD and report 4 HDD

  * (defined as 5 standard drinks per day for men and 4 standard drinks per day for women) in prior 30-days
* 2) enrolled in VA primary care
* 3) planning to initiate MAUD, as determined by a medication order
* 4) between ages 18-80
* 5) willing to be randomized
* 6) Android or iPhone smartphone owners

Exclusion Criteria:

* 1) past 30-day participation in VA or non-VA SUD treatment
* 2) prior episode of MAUD receipt in the last 30 days (initiation of a new episode of MAUD in the 7 days prior to screening allowed)
* 3) plans to be or are pregnant
* 4) severe psychiatric symptoms or psychosocial instability likely to prevent participation in the study protocol, as determined by the referring provider. Veterans aged >80 were excluded because ownership and use of mHealth apps decreases with advancing age. Participants who enter SUD specialty care following randomization will be allowed to continue in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Percent Heavy Drinking Days | 6 months post-baseline
  Change from baseline to 6-month follow-up in percent heavy drinking days (HDD), defined as >4 drinks per day for women and >5 drinks per day for men, was selected as the primary outcome as it combines both frequency and intensity of drinking and is a clinically meaningful measure of change. HDD will be generated from the Timeline Follow Back (TLFB), a retrospective, calendar-based measure that provides information on quantity/frequency of alcohol use in the past 30 days. Percent HDD will be calculated by dividing the number of HDD during a one-month period by 30 days.
Semi-structured qualitative interview data from patients, providers, clinical leaders | 3 months post-baseline
  [Qualitative] Patient, provider, and clinical leader perspectives regarding barriers and facilitators to adoption, implementation, and sustainability of the Stand Down mobile application in combination with medications for AUD in primary care.

SECONDARY OUTCOMES:
Change in Short Inventory of Problems - Revised version (SIP-R) | 6 months post-baseline
  Change from baseline to 6-month follow-up in the Short Inventory of Problems - Revised version (SIP-R), a 17-item questionnaire used to assess negative consequences from drinking. Items are rated on a 4-pt scale (0=Never, 1= Once or a Few Times, 2 = Once or Twice a Week, 3 = Daily or Almost Daily), which yields a total score. Higher scores reflect greater severity of alcohol-related problems.
Change in World Health Organization (WHO) Risk Levels | 6 months post-baseline
  Change from baseline to 6-month follow-up in WHO risk levels, which are defined by average grams of alcohol consumed per day as calculated for each participant from the Timeline Follow Back (TLFB), a retrospective, calendar-based measure that provides information on quantity/frequency of alcohol use in the past 30 days. Participants are categorized into five levels: abstinent (0 g of alcohol/day), low risk (1-40 g/1-20 g of alcohol/day), medium risk (41-60 g/21-40 g of alcohol/day), high risk (61-100 g/41-60 g of alcohol/day), and very high risk (>101 g/>61 g of alcohol/day), with 14g of alcohol being equivalent to 1 standard drink. Reductions in WHO risk levels have been associated with significant improvements in liver function, AUD severity, and functioning among persons with AUD. WHO risk levels are reported as the percentage of participants in each study group representing each risk level.
Change in Client Satisfaction Questionnaire (CSQ) Scores | 6 months post-baseline
  Change from baseline to 6-month follow-up in the Client Satisfaction Questionnaire (CSQ), an 8-item questionnaire used to assess patient satisfaction with substance use treatment. Total scores range from 8 to 32, with higher scores indicating greater satisfaction.
Change in Patient Health Questionnaire Depression Screen (PHQ-9) Scores | 6 months post-baseline
  Change from baseline to 6-month follow-up in the PHQ-9, a 9-item instrument used to screen, diagnose, and monitor the severity of depression. Each item is rated on a 4-point scale (0=Not at all; 1=Several days; 2=More than half the days; and 3=Nearly every day). The total score can range from 0 to 27, with higher scores indicating greater severity of depression.
Change in PTSD Checklist for DSM-5 (PCL-5) Scores | 6 months post-baseline
  Change from baseline to 6-month follow-up in the PTSD Checklist for DSM-5 (PCL-5), a 20-item instrument used to measure presence and severity of PTSD symptoms. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. Each item is rated on a 5-point scale (0= Not at all; 1= A little bit; 2= Moderately; 3= Quite a bit; and 4= Extremely). The total score can range from 0 to 80, with higher scores indicating greater severity of PTSD.
Change in Veterans RAND 12 Item Health Survey Scores | 6 months post-baseline
  Change from baseline to 6-month follow-up in the Veterans RAND 12 Item Health Survey, a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Change in Percent Heavy Drinking Days | 12-months post-baseline
  Change from baseline to 12-month follow-up in in percent HDD, defined as >4 drinks per day for women and >5 drinks per day for men, was selected as the primary outcome as it combines both frequency and intensity of drinking and is a clinically meaningful measure of change. HDD will be generated from the Timeline Follow Back (TLFB), a retrospective, calendar-based measure that provides information on quantity/frequency of alcohol use in the past 30 days. Percent HDD will be calculated by dividing the number of HDD during a one-month period by 30 days.
Change in Short Inventory of Problems - Revised version (SIP-R) | 12-months post-baseline
  Change from baseline to 12-month follow-up in the Short Inventory of Problems - Revised version (SIP-R), a 17-item questionnaire used to assess negative consequences from drinking. Items are rated on a 4-pt scale (0=Never, 1= Once or a Few Times, 2 = Once or Twice a Week, 3 = Daily or Almost Daily), which yields a total score. Higher scores reflect greater severity of alcohol-related problems.
Change in World Health Organization (WHO) Risk Levels | 12-months post-baseline
  Change from baseline to 12-month follow-up in WHO risk levels, which are defined by average grams of alcohol consumed per day as calculated for each participant from the Timeline Follow Back (TLFB), a retrospective, calendar-based measure that provides information on quantity/frequency of alcohol use in the past 30 days. Participants are categorized into five levels: abstinent (0 g of alcohol/day), low risk (1-40 g/1-20 g of alcohol/day), medium risk (41-60 g/21-40 g of alcohol/day), high risk (61-100 g/41-60 g of alcohol/day), and very high risk (>101 g/>61 g of alcohol/day), with 14g of alcohol being equivalent to 1 standard drink. Reductions in WHO risk levels have been associated with significant improvements in liver function, AUD severity, and functioning among persons with AUD. WHO risk levels are reported as the percentage of participants in each study group representing each risk level.
Change in Patient Health Questionnaire Depression Screen (PHQ-9) Scores | 12-months post-baseline
  Change from baseline to 12-month follow-up in the PHQ-9, a 9-item instrument used to screen, diagnose, and monitor the severity of depression. Each item is rated on a 4-point scale (0=Not at all; 1=Several days; 2=More than half the days; and 3=Nearly every day). The total score can range from 0 to 27, with higher scores indicating greater severity of depression.
Number of Participants Receiving VA Outpatient Substance Use Disorder Treatment | 12-months post-baseline
  The total number of participants who received VA outpatient substance use disorder treatment as assessed from visits documented in the VA electronic health record data.
Number of Participants Receiving VA Emergency Department Services | 12-months post-baseline
  The total number of participants who received VA emergency department services as assessed from visits documented in the VA electronic health record data.
Change in PTSD Checklist for DSM-5 (PCL-5) Scores | 12-months post-baseline
  Change from baseline to 12-month follow-up in the PTSD Checklist for DSM-5 (PCL-5), a 20-item instrument used to measure presence and severity of PTSD symptoms. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. Each item is rated on a 5-point scale (0= Not at all; 1= A little bit; 2= Moderately; 3= Quite a bit; and 4= Extremely). The total score can range from 0 to 80, with higher scores indicating greater severity of PTSD.
Change in Veterans RAND 12 Item Health Survey Scores | 12-months post-baseline
  Change from baseline to 12-month follow-up in the Veterans RAND 12 Item Health Survey, a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Hawkins, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (15):
- United States (15):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Veterans Health Care System of the Ozarks, Fayetteville, AR, Fayetteville, Arkansas
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Carl Vinson VA Medical Center, Dublin, GA, Dublin, Georgia
  - Battle Creek VA Medical Center, Battle Creek, MI, Battle Creek, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Richmond VA Medical Center, Richmond, VA, Richmond, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No